CLINICAL TRIAL: NCT01085058
Title: Predictive Value of the "Cytocapacity Test" Following a Single-dose of rHu-G-CSF in Patients With Lymphoproliferative Diseases and High-dose Therapy
Brief Title: Predictive Value of the "Cytocapacity Test" Patients With Lymphoproliferative Diseases and High-dose Therapy
Acronym: CU01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Chugai Pharma GmbH (Unknown)
Responsible Party: Dr. Christian Straka, Univ. of Munich (LMU)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WISP_CU01
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Hodgkin's Disease; Non-Hodgkin Lymphomas; Multiple Myelomas
Keywords: Lymphoproliferative diseases (Hodgkin's disease, non-Hodgkin's lymphomas, multiple myelomas) and high-dose therapy
MeSH Terms: conditions — Hodgkin Disease; Multiple Myeloma | interventions — Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: lenograstim (Experimental): total group
  Interventions: Drug: lenograstim

INTERVENTIONS:
Drug: lenograstim

SUMMARY:
This investigator initiated trial was a prospective, open, single-arm, diagnostic-prognostic study. Patients who received high-dose therapy with autologous stem cell transplantation for the treatment of their lymphoproliferative disease were included into the study.

After completion of the high-dose therapy (day -2 with respect to the stem cell transplantation) the first blood sample A for the cytocapacity test with determination of leukocytes and neutrophils was taken in the evening of day -1. Directly thereafter the study medication was administered. The second blood sample B for the cytocapacity test with determination of leukocytes and neutrophils was taken in the morning of day 0, 12-14 hours after administration of the study medication. Thereafter the stem cell re-infusion was performed.

The primary objective of this study was to show that the cytocapacity test with lenograstim is a useful predictive tool with respect to the risk of post-transplant complications and prolonged myelosuppression, typically occurring after high-dose chemotherapy.

The primary variables were:

* the rate of patients with documented infections
* the time to platelet engraftment

ELIGIBILITY:
Inclusion Criteria:

* Presence of histologically proven lymphoproliferative disease specified as Hodgkin's disease, non-Hodgkin's lymphoma (NHL) or multiple myeloma
* Indication of high-dose therapy and autologous peripheral blood stem cell transplantation
* Availability of a sufficient amount of blood stem cells (CD34+ cells >= 2.0 x 106/kg)
* Age between 18 and 70 years
* High-dose therapy with one of the following high-dose regimes: Melphalan 140 mg/m2 or 200 mg/m2, BEAM, BEAC, BUCY or CBV (the last permitted according to amendment 2, see Section 9.8.1)
* Patient's written consent to participation in this trial

Exclusion Criteria:

* Previous high-dose therapy and blood stem cell transplantation except for melphalan 140 mg/m2 or 200 mg/m2 in patients with multiple myeloma who did not participate in the cytocapacity test previously (according to amendment 2, see Section 9.8.1).
* Known intolerance to lenograstim
* Out-patient therapy following high-dose therapy and blood stem cell transplantation
* Myocardial infarction < 6 months prior to inclusion into the study
* Cardiac arrhythmias Lown IV b
* Clinically manifest cardiac insufficiency (> NYHA II)
* Renal insufficiency with serum creatinine > 2 mg%
* Hepatic diseases with elevated levels of transaminases and bilirubin greater than 3-fold above normal
* Severe infections (HIV, Hepatitis B/C)
* Severe psychiatric diseases
* Non-curative treatment of other malignoma within the past 5 years
* Pregnant women or women breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Incidence of infections
Time to platelet engraftment

REFERENCES:
- [Derived] Straka C, Sandherr M, Salwender H, Wandt H, Metzner B, Hubel K, Silling G, Hentrich M, Franke D, Schwerdtfeger R, Freund M, Sezer O, Giagounidis A, Ehninger G, Grimminger W, Engert A, Schlimok G, Scheid C, Hellmann P, Heinisch H, Einsele H, Hinke A, Emmerich B. Testing G-CSF responsiveness predicts the individual susceptibility to infection and consecutive treatment in recipients of high-dose chemotherapy. Blood. 2011 Feb 17;117(7):2121-8. doi: 10.1182/blood-2010-06-290080. Epub 2010 Dec 16. PMID 21163927